CLINICAL TRIAL: NCT00862589
Title: GLP-1 Suppression of Alpha Cell Secretion in T2DM
Brief Title: Glucagon-Like Peptide-1 (GLP-1) Suppression of Alpha Cell Secretion in Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Kristine Hare/MD, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: H-KA-20070023
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Last update posted 2009-03-18 (Estimated); Status verified 2009-03

CONDITIONS: Hyperglycemia; Hyperglucagonemia; Glucose Intolerance
Keywords: glucagon; GLP-1; hyperglycemia
MeSH Terms: conditions — Hyperglycemia; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: GLP-1 infusion — physiological effect of GLP-1

SUMMARY:
The incretin hormone glucagon-like peptide-1 (GLP-1) has known insulinotrophic and glucagonostatic properties. However, inpatients with type 2 diabetes mellitus (T2DM)it is shown, that the beta cell sensitivity towards GLP-1 is decreased, when comparing to healthy controls. Further, these patients have decreased GLP-1 response to a meal.

The aim of this study is to elucidate if the diabetic hyperglucagonemia, seen in these patients both during fasting and in a postprandial condition, is coursed by a decreased sensitivity to GLP-1 in the diabetic alpha cell.

Ten T2DM patients and ten matched healthy control subjects will be examined on two separate days. Day 1: increasing GLP-1 infusions and Day 2: saline. During both days plasma glucose (PG) will be clamped at fasting level (FPG).

Patients with T2DM will be submitted til a Day 3, here PG will be normalized over-night by an adjustable insulin infusion, on the following day the GLP-1 infusion of Day 1 will be repeated.

The hypothesis is that these patients have decreased alpha cell sensitivity to GLP-1 as is the case with the beta cell sensitivity. This decreased sensitivity, the investigators speculate, contributes the defect suppression og glucagon and thereby to the increased PG levels seen in T2DM. Further the investigators will elucidate if this sensitivity can be increased by normalizing the diabetic PG to a normal FPG level.

ELIGIBILITY:
Inclusion Criteria:

* T2DM according to WHO criteria
* Written consent
* Age > 18 years

Exclusion Criteria:

* Kidney or hepatic disease
* Treatment with insulin or glitazone

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
glucagon suppression

REFERENCES:
- [Derived] Hare KJ, Knop FK, Asmar M, Madsbad S, Deacon CF, Holst JJ, Vilsboll T. Preserved inhibitory potency of GLP-1 on glucagon secretion in type 2 diabetes mellitus. J Clin Endocrinol Metab. 2009 Dec;94(12):4679-87. doi: 10.1210/jc.2009-0921. Epub 2009 Oct 16. PMID 19837930